CLINICAL TRIAL: NCT02477787
Title: Randomized Comparative Study for Efficacy and Safety Evaluation of HLA-haploidentical Hematopoietic Cell Transplantation With or Without Post-transplant Allogeneic Donor-derived Natural Killer Cell Infusion in High-risk Acute Myelogenous Leukemia and Myelodysplastic Syndrome
Brief Title: Randomized Study of Haploidentical Hct and Subsequent Donor nk Cell Infusion in High-risk AML and MDS
Acronym: DNKI-4
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: upon recommendation from the Data Monitoring Committee
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Kyoo-Hyung Lee, MD, PROFESSOR, HEMATOLOGY, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-1091
Record Dates: First submitted 2015-06-11; First posted 2015-06-23 (Estimated); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Acute Myelogenous Leukemia
Keywords: HLA-haploidentical hematopoietic cell transplantation; natural killer cells
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- treatment (Experimental): patients will receive donor-derived NK cell infusion after haploidentical HCT
  Interventions: Biological: allogeneic, donor-derived NK cells
- control (No Intervention): patients will undergo haploidentical HCT but not receive donor-derived NK cells after HCT

INTERVENTIONS:
Biological: allogeneic, donor-derived NK cells — Patients in the study arm will receive donor NK cell infusion around days 13 and 20. A permissible range of infusion time will be +/- 3 days.
  For DNKI to be given on day 13 (DNKI-1), the cell dose is 1-2 x108/kg or about the half of amount generated. For DNKI to be given on day 20 (DNKI-2), the cell dose is up to 5x108/kg.
  Avil 1 ampoule will be given intravenously 30 minutes prior to each NK cell infusions.
  Arms: treatment

SUMMARY:
This is a single center, open label, random comparison phase 2b study. The primary objective of this study is, by random comparison, to assess the anti-leukemia effect of allogeneic, donor-derived natural killer (NK) cells infused after HLA-haploidentical hematopoietic cell transplantation (HCT) in patients with refractory acute myelogenous leukemia (AML).

The secondary objectives of the study are to assess the side effects of donor NK cell infusion, effects of donor NK cell infusion upon HCT outcomes, as well as effects upon post-HCT immune recovery.

DETAILED DESCRIPTION:
5.0 Study design

5.1. Study patient should be enrolled by PI Kyoo-Hyung Lee, MD or Young-Shin Lee, RN.

5.2. Random assignment 5.2.1. Patients were randomly assigned to study arms the day before initiation of conditioning therapy (day -8).

5.2.2. Stratification Refractory AML Stratification 1: Primary refractory vs. relapse-refractory/2 or more relapse Stratification 2: peripheral blood blast <5% vs. ≥5% 5.2.3. extra leukapheresis will be performed form donors assigned to treatment cohort.

High-risk AML Stratification: AML in CR1 with high-risk features vs. AML CR2

High-risk myelodysplastic syndrome (MDS) IPSS intermediate-2 risk vs. IPSS high-risk

6.0. Patient Eligibility

6.1. Patients with refractory AML Refractory AML is defined as follows;

1. Primary refractory: failure to achieve complete remission (CR) after 2 cycles of induction chemotherapy; or, in patient ≥65 years of age, progressive AML after treatment with hypomethylating agent (increase in peripheral blood blast by 50% or increase in bone marrow blast by 25%)
2. Relapse then refractory: recurrence of AML, which is refractory to standard salvage chemo therapy; or, in patient ≥65 years of age, to hypomethylating agent
3. AML in ≥2 relapses

6.2. Patients in AML CR1 with high-risk chromosomal features such as complex abnormality (3 or more abnormalities), -5, 5q-, -7, 7q-, 11q32 abn (non t(9;11)), inv(3), t(3;3), t(6;9), t(9;22), or monosomal karyotype of 2 abnormalites or Patients in AML CR2

6.3 Patients with MDS, in intermediate-2 or high risk categories by IPSS classification

6.4. Patients should be 19 years of age or older

6.5. Patients should have Karnofsky performance scale ≥70

6.6. Patients and cell donors must understand fully and sign informed consent forms

Exclusion

6.7. Pregnant or lactating women

6.8. Patient with abnormal liver function (total bilirubin ≥ 5.0 mg/dl, AST ≥ 5 times upper normal limits)

6.9. Patients with abnormal renal function (creatinine ≥ 3.0 mg/dl)

6.10. Patients with clinically-evident cardiac or pulmonary dysfunction

6.11. Patients with infection that is progressive despite appropriate anti-microbial treatment

6.12 Patients with hypersensitivity to gentamicin

6.13. Patients who had received allogeneic cell therapy

7.0.Treatment Plan

7.1. For the study group of patients, donor NK cells will be generated from the hematopoietic cells. Donor NK cell will be produced in the GCP laboratory at Asan Institute of Life Science by a team of Stem Cell Research Center, Korea Research Institute of Bioscience and Biotechnology.

7.2. Patients will have a triple-lumen Hickman central-venous catheter (CVC) placed. Chest X-ray should be taken after CVC placement to confirm the location and the absence of hematoma formation or pneumothorax.

7.3. Lumbar puncture will be done and preservative free methotrexate 10 mg/m2 (not to exceed 15 mg total) will be given intrathecally.

7.4. Menstruating women will be given norethindrone (Norlutate) 10 mg po daily.

7.5. The preparative regimen (Bu-Flu-ATG; also see Appendix V): 7.5.1. Busulfex (Bu) 3.2 mg/kg/day iv daily on days -7 and -6. Patients who are older than 64 years of age or who have significant co-morbidities may receive Bu on day -7 only.

7.5.2. Fludarabine (Flu) 30 mg/m2/day in D5W 100 ml iv over 30 minutes starting at 4 pm daily on days -7, -6, -5, -4, -3, and -2.

7.5.3. Methylprednisolone 2 mg/kg in D5W 100 ml iv over 30 minutes on days -4, -3, -2, and -1.

7.5.4. Anti-thymocyte globulin (Thymoglobulin, Genzyme Transplant, Cambridge, MA, USA) 2.5 mg/kg/day in N/S 500-800 ml (less than 4 mg/ml) iv over 4 hours starting at 8 am daily on days -3, -2, and -1.

7.6. Hematopoietic stem cell collection from the donors. 7.6.1. The HLA-haploidentical family donor will receive granulocyte colony-stimulating factor (G-CSF, Grasin) 10 ug/kg by subcutaneous (sc) injection for 5 days (from day -3 to day 1). Daily CBC will be done. On days 0, 1, and 2, peripheral blood mononuclear cells will be collected by leukapheresis (Amicus, Fenwal). A female donor or one with poor peripheral vein may have a Quinton or Groshong catheter placed. A sample will be taken for cell count of total cells, mononuclear cells, CD34+ cells, CD3+ cells, CD4+ cells, and CD8+ cells. Cells collected on days 0 and 1, will be transplanted to the patients on the same day without further manipulation. At least 2x106/kg of CD34+ cells should be collected on day 0. If not, additional collection may be scheduled under the discretion of attending physician. G-CSF is the most commonly administered agent to donors for cell-collection and there has been no documented long-term side effect document during last 25 years' use. However, the cell donors in the study will be monitored for possible side effect of G-CSF.

7.6.2. Cell collected on collected on day 2 will be transported to the GCP laboratory for the generation of NK cells (study arm). For details of donor NK cell generation, please see appendix V.

7.7. Peripheral blood hematopoietic cell infusion for transplantation (days 0 or 0-1 or 0-2).

7.7.1. For ABO matched or minor mismatched transplantation, premedication with Avil 45.5 mg iv push and acetaminophen 600 mg po will be given. Stem cells will be infused via CVC over 1 hour.

7.7.2 For major ABO mismatched transplantation, premedication with Avil 45.5 mg iv push, acetaminophen 600 mg po, 10% mannitol 100 g iv over 4 hours beginning 30 minutes before stem cell infusion, and hydrocortisone 250 mg iv immediately before and 30 minutes of stem cell infusion will be given. Stem cells will be infused via CVC over 1 hour.

Donor NK cell infusion (see appendix V) 7.8. The patients in the study arm will receive donor NK cell infusion around days 13 and 20. A permissible range of infusion time will be +/- 3 days.

7.9. For DNKI to be given on day 13 (DNKI-1), the cell dose is 1-2 x108/kg or about the half of amount generated. For DNKI to be given on day 20 (DNKI-2), the cell dose is up to 5x108/kg. 7.10. Avil 1 ampoule will be given intravenously 30 minutes prior to each NK cell infusions.

8.0 Supportive cares. 8.1. Dilantin 15 mg/kg (ABW) in NS 200 ml iv over 1 hour for loading on day -8, then 200 mg po bid through day -6 or -5.

8.2. Clotrimazole powder to groin, axilla, and perianal area bid from day -8 until absolute neutrophil count (ANC) > 3,000/ul.

8.3. Sodium bicarbonate/saline mouthwash qid until mucositis is resolved. 8.4.. Micafungin 50 mg iv qd from Day 1 to ANC > 3,000/ul. 8.5. Ciprofloxacin 500 mg po bid (for selective bowel decontamination) until ANC > 3,000/ul. With the first fever spike, ciprofloxacin is discontinued and broad spectrum antibiotics are begun.

8.6. Acyclovir 250 mg/m2 iv twice a day will be given from day 1, and will be changed into acyclovir 400 mg po bid until the discontinuation of cyclosporine administration.

8.7. G-CSF 450ug iv daily from day 5 to ANC >3,000/ul. 8.8. The patients are hydrated with 0.9 % NS at 100 ml/hr while the patients are receiving busulfan.

8.9. Azithromycin 125 mg iv or po daily starting when ANC >500/ul until 1 year if there is no evidence of GVHD. In patients with GVHD, azithromycin will be continued until resolution of GVHD and discontinuation of immunosuppressive therapy.

8.10. Bactrim 2 t po once a day three times a week when ANC >3,000/ul. 8.11. Intravenous immunoglobulin 500 mg/kg (ABW) iv over 6 hours every 2 weeks starting day 7 until day 90 then monthly until day 180.

9. GVHD prophylaxis 9.1. Cyclosporine 1.5 mg/kg in N/S 100 ml iv over 2-4 hours q12 hrs beginning day -1. Adjust cyclosporine dose to provide appropriate blood level (100-300 ng/ml in whole blood) and according to the change of renal function.

9.2. Cyclosporine dosing will be changed to oral dosing when oral feeding became feasible. Provided that there is no GVHD, cyclosporine dose will be tapered by 10%-20% every 2-4 weeks starting between days 30 and 60 of HCT.

9.3. Cytomegalovirus (CMV) and Epstein-Barr virus (EBV) monitoring: Blood CMV antigenemia assay and quantitative EBV PCR will be done at least weekly starting day -7 until day 100. If CMV antigenemia is positive, preemptive treatment with ganciclovir will be considered as follows; 5 mg/kg iv (every 12 hours for 7 days then) once daily until 1-2 weeks after the negative conversion of CMV antigenemia. When EBV DNA is detected by PCR, infusion of rituximab 375 mg/m2 will be considered weekly until the DNA is no longer detectable.

9.4. CNS prophylaxis: Preservative-free methotrexate will be administered intrathecally after the patient recovered platelet count to over 50,000/mcl. Methotrexate 10 mg/m2 (not to exceed 15 mg total) will be given intrathecally once every 2 weeks for three times (total four doses including one given before preparatory regimen).

10.0. Treatment Evaluation

10.1. Donor work up will include HLA-A, -B, -C, and -DRB1 typing based on PCR-sequencing methods, ABO/Rh typing, CBC with reticulocyte count, chemistry, BUN/phosphorus, electrolytes, coagulation battery, urinalysis with microscopy, EKG, chest PA and lateral, HBsAg, HBsAb, HCV Ab, HIV Ab, VDRL, CMV(IgG), HSV(IgG), EBV serology, Toxoplasma titer (IgG), VZV (IgG) (Appendix II).

10.2. Patient work up will include; HLA-A, -B, -C, and -DRB1 typing based on PCR-sequencing methods, ABO/Rh typing, CBC with reticulocyte count, chemistry, BUN/phosphorus, electrolytes, coagulation battery, urinalysis with microscopy, MUGA scan or echocardiogram, dental consult and Panorex films, ENT consult and PNS films, PFT with DLCO, Chest X-ray, EKG, diagnostic lumbar puncture with fluid battery (cell count, glucose, protein, LD, fungal and bacterial cultures, cytospin), bone marrow aspirate and biopsy with cytogenetics and appropriate molecular tests (such as bcr-abl, pml-rara, aml1-eto), HBsAg, HBsAb, HBcAb (IgG), HCV Ab, HIV Ab, VDRL, CMV (IgG, IgM), HSV (IgG, IgM), EBV serology, Toxoplasma titer (IgG), VZV (IgG), serum pregnancy test (beta-hCG) in females, and isoagglutinin titers if ABO mismatched HCT.

10.3. The status of mixed chimerism will be evaluated by PCR analysis of short tandem repeats (STRs) by multiplex primers. The chimerism status will be analyzed from whole blood DNA after 1, 3, and 6 months after HCT.

10.4. Blood cytomegalovirus (CMV) antigenemia and quantitative EBV PCR assays will be done at least weekly until day 100 of HCT.

10.5. Immune recovery of the patients after stem cell transplantation will be monitored by lymphocyte subset count (Appendix VII) and measurement of Ig G, Ig M, Ig A levels and Ig G subset (G1, G2, G3) on 1, 3, 6, and 12 months after HCT.

10.6. The patients will be followed with physical examination and appropriate blood test including CBC at least every 3 months for 3 years after transplantation and then yearly thereafter.

10.7. Bone marrow examination with cytogenetics will be done 3 to 4 weeks after HCT and, subsequently, as deemed necessary.

10.8. 5 ml of bone marrow and 15 ml of heparinized blood obtained on day -8 will be sent to Asan-KRIBB laboratory for immune phenotyping and functional analysis. In addition, 15 ml of heparinized blood obtained 1, 3, 6, and 12 months after HCT will be sent to Asan-KRIBB laboratory for immune phenotyping and functional analysis (see Appendices VII and VIII).

10.9.Plasma cytokine (interferon-γ, TNF-α, IL-6, IL-15, soluble IL-2 receptor) levels will be measured at 1, 3, 6, and 12 months after HCT.

10.10. On the day of DNKI (days 13 and 20), 5 ml of heparinized peripheral blood will be sent to Asan-KRIBB laboratory for ATG titer determination.

10.11. 96 assessable patients will be enrolled (48 in DNKI arm; 48 in control arm). After enrollment of 40 patients, interim analysis will be performed.

10.12. The enrollment period is 60 months from the approval from Korean Ministry of Food and Drug Safety.

10.13. Continuous variables will be compared using T-test or Mann-Whitney test. Categorical variables will be compared using chi-square test. Lastly, time-event variables will be compared using log-rank test with optional multivariate analysis if necessary.

10.14. Patients will be removed from the study immediately, if the patient withdraws the consent to participate in the study.

11.0. Definition of Endpoints and Response

11.1.The occurrence and severity of side effects of NK cell infusion observed in the study will be monitored and graded according to the Common Toxicity Criteria v3.0(2006; National Cancer Institute). GVHD will be diagnosed and graded by published criteria listed in Appendix III. TRM will be defined as any death occurring after the transplantation without leukemia progression.

11.2.CR is defined as blast less than 5% in the marrow with recovery of neutrophil count over 1,000/ul and no extramedullary disease. CRmarrow is defined as blast less than 5% in the marrow, no blast in the peripheral blood, neutrophil count over 500/ul, platelet count over 20,000/ul, and no extramedullary disease.

11.3.Leukemia recurrence is defined as over 5% leukemia blasts in a bone marrow sample after a previously documented CR. In patients with persistent leukemia after HCT, the day of leukemia progression was defined as the day on which leukemia blasts reappeared in peripheral blood with bone marrow examination showing over 5% persistent blasts.

11.4. Event-free survival will be measured from the day of HCT to leukemia recurrence, transplantation-related mortality, or the last follow-up. Overall survival will be measured from the HCT to death from any cause or the last follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients with refractory AML Refractory AML is defined as follows;

  1. Primary refractory: failure to achieve complete remission (CR) after 2 cycles of induction chemotherapy; or, in patient ≥65 years of age, progressive AML after treatment with hypomethylating agent (increase in peripheral blood blast by 50% or increase in bone marrow blast by 25%)
  2. Relapse then refractory: recurrence of AML, which is refractory to standard salvage chemo therapy; or, in patient ≥65 years of age, to hypomethylating agent
  3. AML in ≥2 relapses
* Patients should be 19 years of age or older
* Patients should have Karnofsky performance scale ≥70
* Patients and cell donors must understand fully and sign informed consent forms

Exclusion Criteria:

* Pregnant or lactating women
* Patient with abnormal liver function (total bilirubin ≥ 5.0 mg/dl, AST ≥ 5 times upper normal limits)
* Patients with abnormal renal function (creatinine ≥ 3.0 mg/dl)
* Patients with clinically-evident cardiac or pulmonary dysfunction
* Patients with infection that is progressive despite appropriate anti-microbial treatment
* Patients with hypersensitivity to gentamicin
* Patients who had received allogeneic cell therapy previously.

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
number of patients who experience progression/recurrence of AML after HCT | up to 60 months

SECONDARY OUTCOMES:
number of patients who achieve engraftment after HCT | up to 6 months
number of patients who develop acute GVHD | up to 4 months
number of patients who develop chronic GVHD | up to 60 months
number of patients who experience donor NK cell infusion-associated toxicity | up to 1 month
number of patients who die after HCT without progression of AML | up to 60 months

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Lee KH, Yoon SR, Gong JR, Choi EJ, Kim HS, Park CJ, Yun SC, Park SY, Jung SJ, Kim H, Lee SY, Jung H, Byun JE, Kim M, Kim SY, Kim JH, Lee JH, Lee JH, Choi Y, Park HS, Lee YS, Kang YA, Jeon M, Woo J, Kang H, Baek S, Kim SM, Kim HM, Cho KH, Choi I. The infusion of ex vivo, interleukin-15 and -21-activated donor NK cells after haploidentical HCT in high-risk AML and MDS patients-a randomized trial. Leukemia. 2023 Apr;37(4):807-819. doi: 10.1038/s41375-023-01849-5. Epub 2023 Mar 17. PMID 36932165